CLINICAL TRIAL: NCT01299168
Title: Multi-centric Observational Study to Analyse the Diagnostic Molecular Features in the Clinical Setting of Kidney Allograft Biopsies
Brief Title: Diagnostic and Therapeutic Applications in Microarrays in Organ Transplantation
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Philip Halloran, Professor, University of Alberta
Other Study IDs: ATAGC-001
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Validation Study of Molecular Diagnostic System; Development of Reporting System for Molecular Diagnosis; Incorporate Molecular Diagnosis Into Diagnostic Standards
Keywords: global gene expression; molecular diagnostic classifiers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Needle kidney biopsy core as per local standard of care
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney Transplant Biopsies for Cause: The study population includes patients with a functioning kidney transplant undergoing a biopsy for clinical indications as standard of care to determine the cause of their graft dysfunction (deterioration in graft function, delayed graft function, proteinuria).

SUMMARY:
The current standard for biopsy-based diagnoses of dysfunction of kidney transplants is the Banff Classification which represents arbitrary international consensus. Recent data-driven approaches using molecular and conventional technologies indicate that mere consensus produces frequently incorrect diagnoses with potential harm to patients due to inappropriate treatment. To address this unmet need and improve diagnostics in the area of organ transplantation, the Alberta Transplant Applied Genomics Centre (ATAGC) has developed a new diagnostic system that combines the molecular and histopathological features of transplant biopsies, plus clinical and laboratory parameters, to create the first Integrated Diagnostic System. The present study will validate and refine this system in 500 prospectively unselected biopsies for clinical indications from American, Canadian and European centres in addition to 300 biopsies already collected. Due to a considerable interest and support from participating Centers, the study is further extended to 1500 prospective biopsies. Thus this is the extension of the INTERCOM study (INTERCOMEX). In addition to demonstrating the feasibility and value of this System in routine patient care and clinical trials, the study will develop and optimize a transparent and user-friendly reporting format to communicate this information to clinicians and obtain detailed feedback on how this system can best improve patient care.

DETAILED DESCRIPTION:
The study has enrolled so far 3012 biopsies from 2313 participants and the results are analyzed for these biopsies. Follow-up data is, and will be collected.

ELIGIBILITY:
Inclusion Criteria:

* All kidney transplant recipients ≥18yrs of age undergoing a kidney biopsy for clinical indications, as determined by their physician or surgeon, will be eligible to enrol in the study.

Exclusion Criteria:

* Patients will be excluded from the study if they decline participation or are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with a functioning kidney transplant undergoing a biopsy for clinicalindications as standard of care to determine the cause of their graft dysfunction (deterioration in graft function, delayed graft function, proteinuria).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-05; Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Validate the Integrated Diagnostic System in the International Collaborative Microarray (INTERCOM) Study | 2013-2016
  1. The rejection classifier predicts Banff diagnosis of any rejection: ABMR, TCMR, or mixed ABMR and TCMR;
  2. The TCMR classifier predicts the presence of Banff TCMR lesions/diagnoses;
  3. The ABMR classifier predicts the presence of ABMR lesions;
  4. In late (>1yr) biopsies for clinical indications, the failure classifier predicts failure within three years.

SECONDARY OUTCOMES:
Demonstrate the feasibility of molecular phenotyping of 300 + 500 kidney transplant biopsies for clinical indications. | 2014-2016
  To test the hypothesis that the molecular phenotype of a newly acquired sample predicts the histologic and clinical features of this sample.
Demonstrate the feasibility of molecular phenotyping of 500 biopsies in real time i.e. returning the molecular phenotyping report in two working days upon sample arrival. | 2015-2016
  Refine the reports based on feedback from the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Philip F Halloran, MD PhD, Principal Investigator — University of Alberta
Locations (26):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Pinnacle Transplant Associates, Harrisburg, Pennsylvania
  - Texas Transplant Institute - Methodist Healthcare System, San Antonio, Texas
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Medical University of Vienna, Vienna, Austria
- Canada (2):
  - Department of Medicine, University of Alberta, Edmonton, Alberta
  - University of British Columbia, St. Paul's Hospital, Vancouver, British Columbia
- University Hospital Merkur, Zagreb, Croatia
- Institute for Experimental and Clinical Medicine (IKEM), Prague, Czechia
- France (2):
  - Hopital Necker, Paris
  - Hopital St. Louis, Paris
- Germany (2):
  - Charité - Universitätmedizin Berlin, Berlin
  - Medizinische Hochschule, Hanover
- Beaumont Hospital, Dublin, Ireland
- Pomeranian Medical University in Szczecin, Szczecin, Poland
- University of Ljubljana, Ljubljana, Slovenia
- Department of Surgery, University of Usan, College of Medicine, Seoul, South Korea
- Vall d'Hebron Hospital, Barcelona, Spain
- University Hospital Zurich, Zurich, Switzerland
- Manchester Royal Infirmary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halloran PF, Famulski KS, Reeve J. Molecular assessment of disease states in kidney transplant biopsy samples. Nat Rev Nephrol. 2016 Sep;12(9):534-48. doi: 10.1038/nrneph.2016.85. Epub 2016 Jun 27. PMID 27345248
- [Background] Halloran PF, Venner JM, Famulski KS. Comprehensive Analysis of Transcript Changes Associated With Allograft Rejection: Combining Universal and Selective Features. Am J Transplant. 2017 Jul;17(7):1754-1769. doi: 10.1111/ajt.14200. Epub 2017 Feb 25. PMID 28101959
- [Background] Halloran PF, Madill-Thomsen KS, Reeve J. The Molecular Phenotype of Kidney Transplants: Insights From the MMDx Project. Transplantation. 2024 Jan 1;108(1):45-71. doi: 10.1097/TP.0000000000004624. Epub 2023 Dec 13. PMID 37310258
- [Background] Madill-Thomsen KS, Halloran PF. Precision diagnostics in transplanted organs using microarray-assessed gene expression: concepts and technical methods of the Molecular Microscope(R) Diagnostic System (MMDx). Clin Sci (Lond). 2024 Jun 5;138(11):663-685. doi: 10.1042/CS20220530. PMID 38819301
- [Background] Halloran PF, Chang J, Mackova M, Madill-Thomsen KS, Akalin E, Alhamad T, Anand S, Arnol M, Baliga R, Banasik M, Blosser CD, Bohmig G, Brennan D, Bromberg J, Budde K, Chamienia A, Chow K, Ciszek M, de Freitas D, Deborska-Materkowska D, Debska-Slizien A, Djamali A, Domanski L, Durlik M, Einecke G, Eskandary F, Fatica R, Francis I, Fryc J, Gill J, Gill J, Glyda M, Gourishankar S, Gryczman M, Gupta G, Hruba P, Hughes P, Jittirat A, Jurekovic Z, Kamal L, Kamel M, Kant S, Kojc N, Konopa J, Lan J, Mannon RB, Matas A, Mazurkiewicz J, Miglinas M, Mueller T, Myslak M, Narins S, Naumnik B, Patel A, Perkowska-Ptasinska A, Picton M, Piecha G, Poggio E, Rajnochova Bloudickova S, Schachtner T, Shojai S, Sikosana ML, Slatinska J, Smykal-Jankowiak K, Solanki A, Veceric Haler Z, Viklicky O, Vucur K, Weir MR, Wiecek A, Wlodarczyk Z, Yang H, Zaky Z, Gauthier PT, Hinze C. A cross-sectional study of the role of epithelial cell injury in kidney transplant outcomes. JCI Insight. 2025 Apr 15;10(10):e188658. doi: 10.1172/jci.insight.188658. eCollection 2025 May 22. PMID 40232852
- [Background] Diebold M, Gauthier PT, Mayer KA, Mackova M, Hinze C, Chang J, Patel UD, Schutz E, Jilma B, Schrezenmeier E, Budde K, Bohmig GA, Halloran PF. Effect of felzartamab on the molecular phenotype of antibody-mediated rejection in kidney transplant biopsies. Nat Med. 2025 May;31(5):1668-1676. doi: 10.1038/s41591-025-03653-3. Epub 2025 Apr 29. PMID 40301559
- [Background] Callemeyn J, Nava-Sedeno JM, Anglicheau D, Beadle J, Brasen JH, Clahsen-van Groningen MC, Cristoferi I, de Loor H, Deutsch A, Essig M, Gwinner W, Halloran PF, Hesselink DA, Koshy P, Kuypers D, Lerut E, Marquet P, Minnee RC, Roufosse C, Sprangers B, Van Craenenbroeck AH, Hatzikirou H, Naesens M. Identification and Cross-Platform Validation of Sparse Molecular Classifiers for Antibody-Mediated and T-Cell-Mediated Rejection After Kidney Transplantation. Kidney Int Rep. 2025 Apr 1;10(6):1806-1818. doi: 10.1016/j.ekir.2025.03.048. eCollection 2025 Jun. PMID 40630324
- [Result] Halloran PF, Pereira AB, Chang J, Matas A, Picton M, De Freitas D, Bromberg J, Seron D, Sellares J, Einecke G, Reeve J. Potential impact of microarray diagnosis of T cell-mediated rejection in kidney transplants: The INTERCOM study. Am J Transplant. 2013 Sep;13(9):2352-63. doi: 10.1111/ajt.12387. Epub 2013 Aug 5. PMID 23915426
- [Result] Halloran PF, Pereira AB, Chang J, Matas A, Picton M, De Freitas D, Bromberg J, Seron D, Sellares J, Einecke G, Reeve J. Microarray diagnosis of antibody-mediated rejection in kidney transplant biopsies: an international prospective study (INTERCOM). Am J Transplant. 2013 Nov;13(11):2865-74. doi: 10.1111/ajt.12465. Epub 2013 Oct 3. PMID 24119109
- [Result] Loupy A, Lefaucheur C, Vernerey D, Chang J, Hidalgo LG, Beuscart T, Verine J, Aubert O, Dubleumortier S, Duong van Huyen JP, Jouven X, Glotz D, Legendre C, Halloran PF. Molecular microscope strategy to improve risk stratification in early antibody-mediated kidney allograft rejection. J Am Soc Nephrol. 2014 Oct;25(10):2267-77. doi: 10.1681/ASN.2013111149. Epub 2014 Apr 3. PMID 24700874
- [Result] Halloran PF, Chang J, Famulski K, Hidalgo LG, Salazar ID, Merino Lopez M, Matas A, Picton M, de Freitas D, Bromberg J, Seron D, Sellares J, Einecke G, Reeve J. Disappearance of T Cell-Mediated Rejection Despite Continued Antibody-Mediated Rejection in Late Kidney Transplant Recipients. J Am Soc Nephrol. 2015 Jul;26(7):1711-20. doi: 10.1681/ASN.2014060588. Epub 2014 Nov 6. PMID 25377077
- [Result] Halloran PF, Merino Lopez M, Barreto Pereira A. Identifying Subphenotypes of Antibody-Mediated Rejection in Kidney Transplants. Am J Transplant. 2016 Mar;16(3):908-20. doi: 10.1111/ajt.13551. Epub 2016 Jan 6. PMID 26743766
- [Result] Reeve J, Chang J, Salazar ID, Lopez MM, Halloran PF. Using Molecular Phenotyping to Guide Improvements in the Histologic Diagnosis of T Cell-Mediated Rejection. Am J Transplant. 2016 Apr;16(4):1183-92. doi: 10.1111/ajt.13572. Epub 2016 Jan 5. PMID 26730747
- [Result] Eskandary F, Bond G, Kozakowski N, Regele H, Marinova L, Wahrmann M, Kikic Z, Haslacher H, Rasoul-Rockenschaub S, Kaltenecker CC, Konig F, Hidalgo LG, Oberbauer R, Halloran PF, Bohmig GA. Diagnostic Contribution of Donor-Specific Antibody Characteristics to Uncover Late Silent Antibody-Mediated Rejection-Results of a Cross-Sectional Screening Study. Transplantation. 2017 Mar;101(3):631-641. doi: 10.1097/TP.0000000000001195. PMID 27120452
- [Result] Aubert O, Loupy A, Hidalgo L, Duong van Huyen JP, Higgins S, Viglietti D, Jouven X, Glotz D, Legendre C, Lefaucheur C, Halloran PF. Antibody-Mediated Rejection Due to Preexisting versus De Novo Donor-Specific Antibodies in Kidney Allograft Recipients. J Am Soc Nephrol. 2017 Jun;28(6):1912-1923. doi: 10.1681/ASN.2016070797. Epub 2017 Mar 2. PMID 28255002
- [Result] Halloran PF, Reeve J, Akalin E, Aubert O, Bohmig GA, Brennan D, Bromberg J, Einecke G, Eskandary F, Gosset C, Duong Van Huyen JP, Gupta G, Lefaucheur C, Malone A, Mannon RB, Seron D, Sellares J, Weir M, Loupy A. Real Time Central Assessment of Kidney Transplant Indication Biopsies by Microarrays: The INTERCOMEX Study. Am J Transplant. 2017 Nov;17(11):2851-2862. doi: 10.1111/ajt.14329. Epub 2017 May 30. PMID 28449409
- [Result] Reeve J, Bohmig GA, Eskandary F, Einecke G, Lefaucheur C, Loupy A, Halloran PF; MMDx-Kidney study group. Assessing rejection-related disease in kidney transplant biopsies based on archetypal analysis of molecular phenotypes. JCI Insight. 2017 Jun 15;2(12):e94197. doi: 10.1172/jci.insight.94197. eCollection 2017 Jun 15. PMID 28614805
- [Result] Madill-Thomsen KS, Wiggins RC, Eskandary F, Bohmig GA, Halloran PF. The Effect of Cortex/Medulla Proportions on Molecular Diagnoses in Kidney Transplant Biopsies: Rejection and Injury Can Be Assessed in Medulla. Am J Transplant. 2017 Aug;17(8):2117-2128. doi: 10.1111/ajt.14233. Epub 2017 Mar 23. PMID 28226404
- [Result] Halloran PF, Matas A, Kasiske BL, Madill-Thomsen KS, Mackova M, Famulski KS. Molecular phenotype of kidney transplant indication biopsies with inflammation in scarred areas. Am J Transplant. 2019 May;19(5):1356-1370. doi: 10.1111/ajt.15178. Epub 2018 Dec 13. PMID 30417539
- [Result] Reeve J, Bohmig GA, Eskandary F, Einecke G, Gupta G, Madill-Thomsen K, Mackova M, Halloran PF; INTERCOMEX MMDx-Kidney Study Group. Generating automated kidney transplant biopsy reports combining molecular measurements with ensembles of machine learning classifiers. Am J Transplant. 2019 Oct;19(10):2719-2731. doi: 10.1111/ajt.15351. Epub 2019 Apr 10. PMID 30868758
- [Result] Madill-Thomsen K, Perkowska-Ptasinska A, Bohmig GA, Eskandary F, Einecke G, Gupta G, Halloran PF; MMDx-Kidney Study Group. Discrepancy analysis comparing molecular and histology diagnoses in kidney transplant biopsies. Am J Transplant. 2020 May;20(5):1341-1350. doi: 10.1111/ajt.15752. Epub 2020 Jan 23. PMID 31846554
- [Result] Einecke G, Reeve J, Gupta G, Bohmig GA, Eskandary F, Bromberg JS, Budde K, Halloran PF; INTERCOMEX investigators. Factors associated with kidney graft survival in pure antibody-mediated rejection at the time of indication biopsy: Importance of parenchymal injury but not disease activity. Am J Transplant. 2021 Apr;21(4):1391-1401. doi: 10.1111/ajt.16161. Epub 2020 Jul 31. PMID 32594646
- [Result] Madill-Thomsen KS, Bohmig GA, Bromberg J, Einecke G, Eskandary F, Gupta G, Myslak M, Viklicky O, Perkowska-Ptasinska A, Solez K, Halloran PF; the INTERCOMEX Investigators. Relating Molecular T Cell-mediated Rejection Activity in Kidney Transplant Biopsies to Time and to Histologic Tubulitis and Atrophy-fibrosis. Transplantation. 2023 May 1;107(5):1102-1114. doi: 10.1097/TP.0000000000004396. Epub 2023 Apr 22. PMID 36575574
- [Result] Halloran PF, Bohmig GA, Bromberg J, Einecke G, Eskandary FA, Gupta G, Myslak M, Viklicky O, Perkowska-Ptasinska A, Madill-Thomsen KS; INTERCOMEX Investigators. Archetypal Analysis of Injury in Kidney Transplant Biopsies Identifies Two Classes of Early AKI. Front Med (Lausanne). 2022 Apr 7;9:817324. doi: 10.3389/fmed.2022.817324. eCollection 2022. PMID 35463013
- [Result] Sikosana MLN, Reeve J, Madill-Thomsen KS, Halloran PF; INTERCOMEX Investigators. Using Regression Equations to Enhance Interpretation of Histology Lesions of Kidney Transplant Rejection. Transplantation. 2024 Feb 1;108(2):445-454. doi: 10.1097/TP.0000000000004783. Epub 2024 Jan 19. PMID 37726883
- [Result] Halloran PF, Madill-Thomsen KS, Bohmig G, Bromberg J, Budde K, Barner M, Mackova M, Chang J, Einecke G, Eskandary F, Gupta G, Myslak M, Viklicky O, Akalin E, Alhamad T, Anand S, Arnol M, Baliga R, Banasik M, Bingaman A, Blosser CD, Brennan D, Chamienia A, Chow K, Ciszek M, de Freitas D, Deborska-Materkowska D, Debska-Slizien A, Djamali A, Domanski L, Durlik M, Fatica R, Francis I, Fryc J, Gill J, Gill J, Glyda M, Gourishankar S, Grenda R, Gryczman M, Hruba P, Hughes P, Jittirat A, Jurekovic Z, Kamal L, Kamel M, Kant S, Kasiske B, Kojc N, Konopa J, Lan J, Mannon R, Matas A, Mazurkiewicz J, Miglinas M, Muller T, Narins S, Naumnik B, Patel A, Perkowska-Ptasinska A, Picton M, Piecha G, Poggio E, Bloudickova SR, Samaniego-Picota M, Schachtner T, Shin S, Shojai S, Sikosana MLN, Slatinska J, Smykal-Jankowiak K, Solanki A, Veceric Haler Z, Vucur K, Weir MR, Wiecek A, Wlodarczyk Z, Yang H, Zaky Z. Subthreshold rejection activity in many kidney transplants currently classified as having no rejection. Am J Transplant. 2025 Jan;25(1):72-87. doi: 10.1016/j.ajt.2024.07.034. Epub 2024 Aug 6. PMID 39117038
- [Result] Hidalgo LG, Madill-Thomsen KS, Reeve J, Mackova M, Gauthier P, Demko Z, Prewett A, Lee M, Alhamad T, Anand S, Arnol M, Baliga R, Banasik M, Blosser CD, Bobba S, Brennan D, Bromberg J, Budde K, Chamienia A, Chow K, Ciszek M, Costa N, Deborska-Materkowska D, Debska-Slizien A, Domanski L, Fatica R, Francis I, Fryc J, Gill J, Gill J, Glyda M, Gourishankar S, Gryczman M, Gupta G, Hruba P, Hughes P, Jittirat A, Jurekovic Z, Kamal L, Kamel M, Kant S, Kojc N, Konopa J, Kumar D, Lan J, Lowe D, Mazurkiewicz J, Miglinas M, Moinuddin I, Mueller T, Myslak M, Naumnik B, Paczek L, Patel A, Perkowska-Ptasinska A, Piecha G, Poggio E, Bloudickova SR, Regele H, Schachtner T, Shojai S, Sikosana MLN, Slatinska J, Smykal-Jankowiak K, Haler ZV, Viklicky O, Vucur K, Weir MR, Wiecek A, Zaky Z, Halloran PF. Improving the histologic detection of donor-specific antibody-negative antibody-mediated rejection in kidney transplants. Am J Transplant. 2025 Aug 23:S1600-6135(25)02943-0. doi: 10.1016/j.ajt.2025.08.029. Online ahead of print. PMID 40854490
- [Derived] Halloran PF, Madill-Thomsen KS, Bohmig GA, Myslak M, Gupta G, Kumar D, Viklicky O, Perkowska-Ptasinska A, Famulski KS; INTERCOMEX Investigators. A 2-fold Approach to Polyoma Virus (BK) Nephropathy in Kidney Transplants: Distinguishing Direct Virus Effects From Cognate T Cell-mediated Inflammation. Transplantation. 2021 Nov 1;105(11):2374-2384. doi: 10.1097/TP.0000000000003884. PMID 34310102
- [Derived] Madill-Thomsen KS, Bohmig GA, Bromberg J, Einecke G, Eskandary F, Gupta G, Hidalgo LG, Myslak M, Viklicky O, Perkowska-Ptasinska A, Halloran PF; INTERCOMEX Investigators. Donor-Specific Antibody Is Associated with Increased Expression of Rejection Transcripts in Renal Transplant Biopsies Classified as No Rejection. J Am Soc Nephrol. 2021 Nov;32(11):2743-2758. doi: 10.1681/ASN.2021040433. Epub 2021 Jul 12. PMID 34253587
- [Derived] Halloran PF. Integrating molecular and histologic interpretation of transplant biopsies. Clin Transplant. 2021 Apr;35(4):e14244. doi: 10.1111/ctr.14244. Epub 2021 Feb 17. No abstract available. PMID 33595110
- [Derived] Halloran PF, Bohmig GA, Bromberg JS, Budde K, Gupta G, Einecke G, Eskandary F, Madill-Thomsen K, Reeve J; INTERCOMEX investigators. Discovering novel injury features in kidney transplant biopsies associated with TCMR and donor aging. Am J Transplant. 2021 May;21(5):1725-1739. doi: 10.1111/ajt.16374. Epub 2020 Nov 30. PMID 33107191
- [Derived] Venner JM, Famulski KS, Reeve J, Chang J, Halloran PF. Relationships among injury, fibrosis, and time in human kidney transplants. JCI Insight. 2016 Jan 21;1(1):e85323. doi: 10.1172/jci.insight.85323. PMID 27699214